CLINICAL TRIAL: NCT06058338
Title: Multi-level Evaluation of Produce Prescription Projects on Type 2 Diabetes-related Outcomes: A Pathway to Policy Change by Addressing Social Determinants of Health
Brief Title: Pathway for Produce Prescriptions in Diabetes Management
Acronym: PPT2D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Gretchen Swanson Center for Nutrition (Other)
Collaborators: American Diabetes Association (Other); University of Colorado, Denver (Other); University of California, San Francisco (Other); Children's Hospital Medical Center, Cincinnati (Other); Lawndale Christian Health Center (Other); Virtua Health (Other); Parkview Hospital, Indiana (Other); Presbyterian Healthcare Services (Unknown); Market Umbrella (Unknown)
Responsible Party: Principal Investigator, Carmen Byker Shanks, Principal Research Scientist, Gretchen Swanson Center for Nutrition
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 7-22-ICTSN-40
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Type 2 Diabetes
Keywords: Produce Prescriptions; Social Determinants of Health; Food Security
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Intervention arm participants will receive produce prescription services for a defined period of time (4-6months)
  Interventions: Behavioral: Produce Prescription
- Control Arm (No Intervention): Control arm participants will not receive produce prescriptions but will receive standard of care services for diabetes management

INTERVENTIONS:
Behavioral: Produce Prescription — Produce prescriptions mitigate health and food access inequities by partnering with healthcare providers to prescribe fruits and vegetables via financial incentives to patients experiencing food insecurity, low income, and/or chronic disease(s) risk.
  Arms: Intervention Arm

SUMMARY:
Fruit and vegetable (FV) intake decrease the risk of type 2 diabetes (T2D) and is important for T2D management but is difficult to achieve in adequate amounts for those with a low- income. Produce Prescription (PPR) projects are an intervention aligned with the social determinants of health that help individuals with a low-income purchase FV by providing an incentive. The impacts of PPR projects on populations with T2D and a low-income is less understood. The Multi-level evaluation of Produce Prescription Projects on type 2 diabetes- related outcomes: A pathway to policy change by addressing social determinants of health study will determine the impact of PPR projects on hemo-globin A1c (HbA1c; primary outcome), fruit and vegetable intake (FVI), food security, and related behaviors among a diverse sample of PPR participants diagnosed with T2D and low-income (Aim 1), and will conduct a cost and cost-effective analysis of PPR projects (Aim 2), and a mixed methods process evaluation to understand feasibility and best practices for PPR projects for people with/at risk for T2D (Aim 3). We hypothesize that PPR participants will see greater declines in HbA1c and improvements in other health and food-related behaviors, compared to the Standard of Care. We will recruit five GusNIP PPR projects, whose healthcare partners serve patients with T2D, and who have participating and matched non-participating control populations. We will collect data at baseline and post-intervention using validated, survey modules, clinical measures, and cost data. Five types of data will be used for this project: 1.Health and healthcare utilization data from the EHR or point-of-care, 2.Participant survey data, 3.Qualitative data, 4.Program cost data (NOT human subjects), and 5.Process data (NOT human subjects). Information extracted from medical records includes HbA1c, weight, and blood pressure and will be collected at 2 time points (months 0,6), following their standard of care protocols. Staff will also extract healthcare utilization data (e.g., #primary care and #ER visits) from the EHR at each of site. Primary analyses will use an intention to treat strategy. Analysis will include a linear mixed-effect model to the HbA1c with an interaction between group and time to examine whether there is a difference in HbA1c trajectories between intervention and control groups. Similar models will be used to determine impact on each of the secondary outcomes (e.g., healthcare utilization, BMI).

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with Type 2 diabetes
2. have clinically screened positive for food insecurity and/or be income-eligible to receive Medicaid and/or SNAP-benefits
3. ≥ 18 years of age, and
4. be a patient at a participating healthcare site.

Exclusion Criteria:

1. people who pregnant or nursing and
2. plans to move away during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | Months 0,6
  Participant HbA1c will be collected by point-of-care venipuncture or from lab draws in electronic medical records.

SECONDARY OUTCOMES:
Body Mass Index | Months 0,6
  Participant BMI will be calculated from height/weight measurements from electronic medical records.
Blood pressure | Months 0,6
  Participant systolic and diastolic blood pressure measurements will be collected from electronic medical records.
Fruit and vegetable intake | Months 0,6
  Participant fruit and vegetable intake as measured by the NCI/NIH Dietary Screener Questionnaire (DSQ) 10-item fruit and vegetable module.
Food security | Months 0,6
  Participant food security status as measured by the USDA 6-item food security survey.
Diabetes distress | Months 0,6
  Participant diabetes distress as measured by the Problem Areas in Diabetes Scale (PAID-5) using the scale of 0, not a problem, to 4, serious problem with higher scores indicating more emotional stress from living with diabetes
Health-related Quality of Life | Months 0,6
  Participant health-related quality of life as measured by the Short Form (SF)-12 module that addresses 8 domains of physical and mental health along a scale ranging from 0 to 100, with higher scores indicating better physical and mental health functioning
Self-efficacy | Months 0,6
  Participant self-efficacy for eating fruits and vegetables as measured by a single survey question using a 5 point scale from 0 to 5 with 0 indicating not at all confident and 5 indicating very confident.
Self-reported health | Months 0,6
  Participant self-reported health status as measured by a single survey question using a 5 point scale from 0 to 5 with 0 indicating poor health and 5 indicating excellent health
Program satisfaction | Month 6
  Participant produce prescription program satisfaction as measured by a single survey question using a 5 point scale from 0 to 5 with 0 indicating very negative satisfaction and 5 indicating very positive satisfaction

OTHER OUTCOMES:
Program cost | Months 1-6
  The estimated cost to operate a produce prescription program for four-to-six months as measured by clinic administrative records and staff interviews.
Cost-effectiveness (HbA1c -1%) | Months 0-6
  The cost-effectiveness of produce prescription program on a 1% decrease in HbA1c over four-to-six months as measured by clinic administrative records and staff interviews (combines outcome 1 and outcome 11).
Cost-effectiveness (HbA1c <7%) | Months 0-6
  The cost-effectiveness of produce prescription program on reducing HbA1c to <7% among participants with HbA1c >=7% as measured by clinic administrative records and staff interviews (combines outcome 1 and outcome 11).
Program reach | Months 1-6
  A process evaluation measure for the proportion of intervention group participants that received at least one produce prescription incentive as measured by clinic administrative records.
Dose delivered | Months 1-6
  A process evaluation measure for the percentage of intended intervention components delivered to participants (e.g., dollar amount and frequency of prescriptions issued) as measured by clinic administrative records.
Dose received | Months 1-6
  A process evaluation measure for the percentage of intended intervention components received by participants (e.g., number of nutrition education activities attended) as measured by clinic administrative records.
Fidelity | Months 1-6
  A process evaluation measure for how well intervention components were delivered according to plan (e.g., number of nutrition educational activities delivered compared to the number scheduled) as measured by clinic administrative records and semi-structured interviews.
Participant experiences | Months 7-8
  A process evaluation measure for participant experience with the produce prescription as measured by participant focus groups.
Program feasibility | Months 1-2, 7-8
  A process evaluation measure for the feasibility of produce prescription programs as measured by interviews with key partners.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Byker Shanks, PhD, Principal Investigator — Gretchen Swanson Center for Nutrition
Locations (5):
- United States (5):
  - Chicago Botanic Gardens - Farm on Ogden, Chicago, Illinois
  - Parkview Hospital, Fort Wayne, Indiana
  - Market Umbrella, New Orleans, Louisiana
  - Virtua Health, Marlton, New Jersey
  - Presbyterian Healthcare Services, Santa Fe, New Mexico